CLINICAL TRIAL: NCT04122833
Title: A Next-generation Sequencing Analysis to Investigate the Clinical Impact of Concomitant Genetic Alterations in the Patients With Advanced EGFR-mutated Lung Adenocarcinoma: A Multicenter Study.
Brief Title: Impact of Concomitant Genetic Alterations in EGFR Mutated Adenocarcinoma by NGS Analysis: A Multicenter Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Konkuk University Medical Center (Other)
Collaborators: Roche Diagnostics GmbH (Industry); Foundation Medicine (Industry)
Responsible Party: Principal Investigator, Kye Young Lee, Professor, Konkuk University Medical Center
Other Study IDs: ML41560
Record Dates: First submitted 2019-10-03; First posted 2019-10-10 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Adenocarcinoma of Lung; EGFR Activating Mutation
Keywords: next generation sequencing
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Next generation sequencing — observational study

SUMMARY:
The concomitant co-mutation with epidermal growth factor receptor (EGFR) mutation might influence the clinical outcomes. The investigators will identify the impact of concommitant mutation on clinical outcome in patients with advanced -EGFR mutated adenocarcinoma.

The investigators will compare the genetic alterations between tumors of pre and post Tyrosin Kinase Inhibitor(TKI) treatments and predict the resistance mechanism for EGFR-TKIs by next-generation sequencing(NGS) analysis.

DETAILED DESCRIPTION:
The current standard therapies in the treatment of advanced EGFR-mutated lung cancer patients are the 1st or 2nd EGFR-TKIs. Although 70-80% of patients treated by EGFR-TKIS show good responses, they have progression after around 12 months. The concomitant co-mutation with EGFR mutation might influence the drug response of EGFR TKI. The investigators will compare the progression-free survival (PFS) of EGFR-TKI according to co-occuring mutations.

The patients experience the change of molecular profiles after using the TKI. Therefore, the investigators will investigate the molecular profiles through NGS panel with foundation medicine in the tissue of pre/post EGFR-TKI, compare the change of the molecular profiles and tumor mutation burden(TMB), and identify novel mechanisms of drug resistance.

The investigators will collect the tumor tissues and blood of around 80 patients in multi-centers prospectively. Then, They will be sent to FoundationOne in the US and perform NGS analysis. The type of EGFR-TKIs would be selected according to physicians' preference. NGS will be performed twice before the EGFR-TKIs treatment and after the progression.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Age ≥19 years
3. EGFR-mutated stage IV lung adenocarcinoma patients
4. Archival biopsy tissues which are from core needle biopsies, endobronchial ultrasound (EBUS) guided- lymph node biopsy or lymph node excisional biopsy at baseline and at radiologic progression
5. Availability of the 10 unstained slides and 1 H&E slides at pre/ post TKI treatment
6. Samples should contain a minimum of 20% viable tumor cells that preserve

Exclusion Criteria:

Tumor tissue from bone metastases that have been decalcified are not acceptable.

-

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: EGFR-mutated stage IV lung adenocarcinoma patients
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of mutation profiles between pre/post TKI treatment | through study completion, an average of 1 year
  Comparison of the kinds of the mutation between pre- and post TKI treatment

SECONDARY OUTCOMES:
PFS according to the co-occurring mutations with pre-TKI treatment | through study completion, an average of 1 year
  The investigators will compared the PFS according to the kinds of co-occuring genetic alteration in patient with EGFR -mutated adenocarcinoma before the EGFR TKI treatment
The number and the kinds of co-occurring mutations on tumors before and after TKI treatment | through study completion, an average of 1 year
  The investigators will collect the information about the number and the kinds of co-occurring mutations on tumors before and after TKI treatment in Foundation medicine NGS
The correlation between the change of variant allele frequency(VAF) and drug response in matched tumors tissues before and after TKI treatment | through study completion, an average of 1 year
  The investigators will analyze the correlation with the change of the VAF and PFS in matched tumors tissues before and after TKI treatment
Tumor mutation burden in tumors tissues before and after TKI treatment | through study completion, an average of 1 year
  The investigators will compare the TMB in tumors tissues before and after TKI
The concordance the the mutation profiles in the NGS results of tissue and blood in the same patients | through study completion, an average of 1 year
  The investigators will compare the concordance of the mutation profile in tumors and blood before TKI treatment

CONTACTS AND LOCATIONS:
Overall Officials: In Ae Kim, MD. Ph.D, Study Director — Kunkuk University Medical Center
Locations (2):
- South Korea (2):
  - Asan medical center, Seoul
  - Catholic university medical center, Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sequist LV, Yang JC, Yamamoto N, O'Byrne K, Hirsh V, Mok T, Geater SL, Orlov S, Tsai CM, Boyer M, Su WC, Bennouna J, Kato T, Gorbunova V, Lee KH, Shah R, Massey D, Zazulina V, Shahidi M, Schuler M. Phase III study of afatinib or cisplatin plus pemetrexed in patients with metastatic lung adenocarcinoma with EGFR mutations. J Clin Oncol. 2013 Sep 20;31(27):3327-34. doi: 10.1200/JCO.2012.44.2806. Epub 2013 Jul 1. PMID 23816960
- [Background] Kim Y, Lee B, Shim JH, Lee SH, Park WY, Choi YL, Sun JM, Ahn JS, Ahn MJ, Park K. Concurrent Genetic Alterations Predict the Progression to Target Therapy in EGFR-Mutated Advanced NSCLC. J Thorac Oncol. 2019 Feb;14(2):193-202. doi: 10.1016/j.jtho.2018.10.150. Epub 2018 Nov 1. PMID 30391576
- [Background] Offin M, Rizvi H, Tenet M, Ni A, Sanchez-Vega F, Li BT, Drilon A, Kris MG, Rudin CM, Schultz N, Arcila ME, Ladanyi M, Riely GJ, Yu H, Hellmann MD. Tumor Mutation Burden and Efficacy of EGFR-Tyrosine Kinase Inhibitors in Patients with EGFR-Mutant Lung Cancers. Clin Cancer Res. 2019 Feb 1;25(3):1063-1069. doi: 10.1158/1078-0432.CCR-18-1102. Epub 2018 Jul 25. PMID 30045933
- [Background] Yu HA, Suzawa K, Jordan E, Zehir A, Ni A, Kim R, Kris MG, Hellmann MD, Li BT, Somwar R, Solit DB, Berger MF, Arcila M, Riely GJ, Ladanyi M. Concurrent Alterations in EGFR-Mutant Lung Cancers Associated with Resistance to EGFR Kinase Inhibitors and Characterization of MTOR as a Mediator of Resistance. Clin Cancer Res. 2018 Jul 1;24(13):3108-3118. doi: 10.1158/1078-0432.CCR-17-2961. Epub 2018 Mar 12. PMID 29530932
- [Background] Socinski MA, Villaruz LC, Ross J. Understanding Mechanisms of Resistance in the Epithelial Growth Factor Receptor in Non-Small Cell Lung Cancer and the Role of Biopsy at Progression. Oncologist. 2017 Jan;22(1):3-11. doi: 10.1634/theoncologist.2016-0285. Epub 2016 Nov 7. PMID 27821794